CLINICAL TRIAL: NCT06699108
Title: A Multi-Center, Randomized, Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of VGR-R01 in Subjects With Bietti Crystalline Dystrophy
Brief Title: Study to Evaluate the Efficacy and Safety of VGR-R01 Gene Therapy in Patients With Bietti Crystalline Dystrophy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGR-R01-301
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Bietti Crystalline Dystrophy; Inherited Retinal Diseases
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental)
  Interventions: Drug: VGR-R01
- Control group (No Intervention)

INTERVENTIONS:
Drug: VGR-R01 — Subretinal injection of VGR-R01 (0.1 mL)
  Arms: interventional group

SUMMARY:
This is a phase 3 study to evaluate the efficacy and safety of VGR-R01 in subjects with Bietti Crystalline Dystrophy.

This is a multicenter, randomized controlled study which will enroll 45 subjects.

DETAILED DESCRIPTION:
VGR-R01 is a novel AAV vector carrying the human CYP4v2 coding sequence. This study is intended to assess the efficacy of VGR-R01 in subjects with Bietti crystalline dystrophy (BCD) based on the change from baseline in best corrected visual acuity (BCVA) of the study eyes.

30 subjects will be enrolled in the intervention group and will receive monocular administration of VGR-R01, and 15 subjects in the control group will not receive any intervention. After completion of the trial, the untreated eyes will receive administration of VGR-R01 in subsequent clinical trial.

ELIGIBILITY:
Key Inclusion Criteria:

1. Able to provide informed consent and comply with requirements of the study;
2. ≥18 years and <70 years of age;
3. Confirmed diagnosis of Bietti Crystalline Dystrophy and molecular diagnosis of CYP4V2 mutations (homozygotes or compound heterozygotes);
4. Hand Motion ≤ BCVA ≤ 60 ETDRS letters in the study eye;

Key Exclusion Criteria:

1. Have insufficient viable retinal photoreceptor cells based on investigator's decision;
2. Have current ocular or periocular infections, or endophthalmitis;
3. Have any significant ocular disease/disorder other than BCD, including age-related macular degeneration, diabetic retinopathy, optic neuropathy, significant lens opacity, glaucoma, uveitis, retinal detachment, etc;
4. Have intraocular surgery history except cataract surgery in the study eye;
5. Have or potentially require of systemic medications that may cause eye injure;
6. Have contraindications for corticosteroids or immunosuppressant;
7. Unwilling or unable to have the planned follow-up;
8. Abnormal coagulation function or other clinically significant abnormal laboratory results;
9. Have malignancies or history of malignancies;
10. History of immunodeficiency (acquired or congenital); Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with change in BCVA in the study eyes of BCD subjects as assessed by ETDRS | Baseline up to Week 52
  Change in the BCVA assessment from screening in the study eye of BCD subjects will be compared to controls

SECONDARY OUTCOMES:
Change from baseline in BCVA | Baseline up to Week 52
  BCVA will be assessed with the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart. Testing Protocol will be followed (confidential). Change in the BCVA assessment from baseline in treated eyes of intervention group will be compared to controls.
Change from baseline in multi-luminance mobility test (MLMT) score of the study eye | Baseline up to Week 52
  Subjects will navigate a standardized mobility maze under set conditions as specified times during the study. The mobility testing will follow a standardized administration and data acquisition protocol and may only be administered by site staff certified in the methodology.
Changes from baseline in Microperimetry indexes | Baseline up to Week 52
  Number of subjects with change in fixation stability or light sensitivity in treated eyes of intervention group will be compared to controls
Change from baseline in optical coherence tomography (OCT) | Baseline up to Week 52
  Change from baseline in central retinal thickness (CRT) as imaged by OCT
Counts, frequencies and percentages of AE, SAE and other safety evaluation | Baseline up to Week 52
  Ocular/non-ocular adverse events are collected. The ophthalmic examination will include BCVA, IOP, slitlamp examination, angiography and SD-OCT, etc. If any potential changes accompanied by clinical symptoms, or results in a change of medical intervention, the findings will be considered as clinically significant based on investigator's decision
Number of subjects with the presence of immunogenicity | Baseline up to Week 52
  Assessed as presence of systemic cell-mediated or humoral responses to capsid or transgene product

OTHER OUTCOMES:
Changes from baseline in visual field index | Baseline up to Week 52
  Assessed by Humphery static visual field testing.
Change from baseline in PRO measures | Baseline up to Week 52
  As assessed by the NEI-VFQ-25 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Vitalgen Biopharma Co.,Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGR-R01 is fully approved